CLINICAL TRIAL: NCT00624169
Title: Peptic Ulcer Perforation Study - an Optimized Perioperative Course for Patients Surgically Treated for Peptic Ulcer Perforation
Brief Title: Peptic Ulcer Perforation Study
Acronym: PULP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Odense University Hospital (Other); Bispebjerg Hospital (Other); Hvidovre University Hospital (Other); Aarhus University Hospital (Other); Hillerod Hospital, Denmark (Other); Helsingør hospital (Unknown)
Responsible Party: Morten Hylander Møller. MD, Department of Anaesthesiology and Intensive Care Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-D-2007-0044
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Peptic Ulcer Perforation
Keywords: Perforated peptic ulcer; Mortality
MeSH Terms: conditions — Peptic Ulcer Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: An optimized perioperative course — A number of interventions before, during and after surgery

SUMMARY:
The objective of this study is to implement an optimized perioperative course for patients surgically treated for peptic ulcer perforation in order to improve the outcome for these patients.

The optimized perioperative course consists of a number of interventions carried out before, during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients surgically treated for benign peptic ulcer perforation

Exclusion Criteria:

* Age < 18 years
* Pregnant and breastfeeding women
* Malign ulcer perforation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
All cause mortality rate | Within 30 days of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bo Belhage, MD, PhD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Bispebjerg; Lars N Jørgensen, MD, PhD, Principal Investigator — Department of Gastrointestinal Surgery, Copenhagen University Hospital Bispebjerg; Iben Rosenberg, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Hillerød; Anders U Neuenschwander, MD, Principal Investigator — Department of Gastrointestinal Surgery, Copenhagen University Hospital Hillerød; Ulf Sigild, MD, Principal Investigator — Department of Gastrointestinal Surgery, Copenhagen University Hospital Helsingør; Anne-Margrete Hedengran, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Helsingør; Peter Holde, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care, Odense University Hospital; Erik Zimmermann-Nielsen, MD, PhD, Principal Investigator — Department of Gastrointestinal Surgery, Odense University Hospital; Anita Lauritsen, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Århus University Hospital; Jørgen Bendix, MD, Principal Investigator — Department of Gastrointestinal Surgery, Århus University Hospital; Sven Adamsen, MD, Principal Investigator — Department of Gastrointestinal Surgery, Copenhagen University Hospital Herlev; Morten H Møller, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Herlev; Ann M Møller, MD, PhD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Herlev; Jens-Ulrik S Jensen, MD, Principal Investigator — Department of Clinical Microbiology / Copenhagen HIV Programme, Copenhagen University Hospital Hvidovre; Niels Fogh-Andersen, MD, Principal Investigator — Department of Clinical Biochemistry, Copenhagen University Hospital Herlev
Locations (7):
- Denmark (7):
  - Århus University Hospital, Aarhus
  - Copenhagen University Hospital Bispebjerg, Copenhagen NV
  - Copenhagen University Hospital Helsingør, Elsinore
  - Copenhagen University Hospital Herlev, Herlev
  - Copenhagen University Hospital Hillerød, Hillerød
  - Copenhagen University Hospital Hvidovre, Hvidovre
  - Odense University Hospital, Odense

REFERENCES:
- [Derived] Moller MH, Vester-Andersen M, Thomsen RW. Long-term mortality following peptic ulcer perforation in the PULP trial. A nationwide follow-up study. Scand J Gastroenterol. 2013 Feb;48(2):168-75. doi: 10.3109/00365521.2012.746393. Epub 2012 Dec 10. PMID 23215900
- [Derived] Moller MH, Adamsen S, Thomsen RW, Moller AM; Peptic Ulcer Perforation (PULP) trial group. Multicentre trial of a perioperative protocol to reduce mortality in patients with peptic ulcer perforation. Br J Surg. 2011 Jun;98(6):802-10. doi: 10.1002/bjs.7429. Epub 2011 Mar 25. PMID 21442610